CLINICAL TRIAL: NCT02711540
Title: Retrospective Analysis of Procedural Aspects of Transcatheter Aortic Valve Implantation (TAVI) on Peri-procedural Stroke Rates in the United Kingdom
Brief Title: Retrospective Analysis of Procedural Aspects of Transcatheter Aortic Valve Implantation (TAVI) on Peri-procedural Stroke
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Sussex County Hospital (Other)
Responsible Party: Principal Investigator, David Hildick-Smith, Consultant Cardiologist, Royal Sussex County Hospital
Other Study IDs: TAVIStrokePredictors
Record Dates: First submitted 2016-03-02; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-TAVI Balloon Aortic Valvuloplasty: This is the cohort of patients in the study who did receive Balloon Aortic Valvuloplasty (BAV) prior to TAVI implantation
  Interventions: Procedure: Balloon Aortic Valvuloplasty
- No Pre-TAVI Balloon Aortic Valvuloplasty: This is the cohort of patients in the study who did not receive Balloon Aortic Valvuloplasty (BAV) prior to TAVI implantation

INTERVENTIONS:
Procedure: Balloon Aortic Valvuloplasty — Some patients receive BAV prior to TAVI implantation to facilitate better deployment of the TAVI valve
  Groups: Pre-TAVI Balloon Aortic Valvuloplasty

SUMMARY:
Retrospective analysis of all patients receiving TAVI in the United Kingdom (UK). Stroke rates following TAVI are roughly 3%. There are several device and procedure related characteristics which may increase the risk of stroke. We will examine if there is a signal in the UK registry. This will be important is TAVI is to be extended down to lower risk patient cohorts.

DETAILED DESCRIPTION:
Retrospective analysis of all patients receiving TAVI in the UK. Stroke rates following TAVI are roughly 3%. There are several device and procedure related characteristics which may increase the risk of stroke. We will examine if there is a signal in the UK registry. This will be important is TAVI is to be extended down to lower risk patient cohorts.

Factors to be examined include (but not limited to):

need for Pre-procedure Balloon aortic Valvuloplasty (BAV) Need for two valves need for post-dilatation need for rapid ventricular burst pacing

ELIGIBILITY:
Inclusion Criteria:

* Had TAVI procedure in UK

Exclusion Criteria:

* Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had TAVI in the UK
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Stroke | 30 days
  Stroke, defined as new neurological deficit with corresponding change on CT scan of brain, is a self reported event following TAVI. All centres performing TAVI in the United Kingdom are required to report this to the National Institute for Cardiovascular Outcomes Research (NICOR) registry which is being analysed in this study

IPD SHARING:
Plan to Share IPD: No